CLINICAL TRIAL: NCT02151383
Title: Multicenter, Open-label, Dose Escalation Study to Evaluate Safety, Tolerability and Pharmacokinetics of RLX030 in Addition to Standard of Care in Pediatric Patients From Birth to <18 Years of Age, Hospitalized With Acute Heart Failure
Brief Title: Pharmacokinetics & Safety of Serelaxin on Top of Standard of Care Therapy in Pediatric Patients With Acute Heart Failure
Acronym: RELAX-PEDS-PK
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated early based on Adult AHF study CRLX030A2301 results
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRLX030A2208; 2013-002847-28 (EudraCT Number)
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Results first posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-05

CONDITIONS: Acute Heart Failure
Keywords: Acute heart failure; RELAX-AHF-PEDIATRIC PK; AHF
MeSH Terms: interventions — serelaxin protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Serelaxin (Experimental): Serelaxin was administered intravenously on top of standard therapy for acute heart failure, for a total of 48 hours.
  Interventions: Drug: Serelaxin

INTERVENTIONS:
Drug: Serelaxin — Serelaxin was administered intravenously for up to 48 hours.
  Other Names: RLX030

SUMMARY:
The purpose of the study was to evaluate the safety, tolerability and pharmacokinetics of an intravenous infusion of serelaxin on top of standard of care therapy, in pediatric patients with acute heart failure (AHF)

DETAILED DESCRIPTION:
The study was terminated early and the pediatric development of serelaxin in the treatment of acute heart failure (AHF) discontinued, following the results of the phase III study RELAX-AHF-2 (CRLX030A2301/NCT01870778) study in adult patients with AHF. Whilst no new safety concerns associated with serelaxin were observed, the study in adults did not meet either of its primary endpoints

ELIGIBILITY:
Key Inclusion criteria:

* Body weight ≥2.5 kg to ≤120 kg
* Hospitalized in an intensive care unit or step-down unit with the following:
* - Signs and symptoms of acute heart failure of any etiology
* - Stable dose of vasoactive and/or inotropic drugs
* - For non-surgical patients echocardiographic evidence of reduced ventricular function (ejection fraction <50% or fractional shortening <28%)
* Systolic blood pressure (SBP) ≥25th percentile SBP for age and gender.

Key Exclusion criteria:

* Moderate to severe left ventricular outflow tract, mitral stenosis, or aortic arch obstruction
* Single ventricle physiology
* Fixed pulmonary hypertension
* Blood lactate levels >5 mmol/L at screening
* Birth < 36 weeks post-conceptual age (for patients <1year old)
* Confirmed or clinically suspected systemic infection or severe localized infection
* Dyspnea or acute lung injury primarily due to non-cardiac causes
* Patients with severe renal impairment, those known to have significant renal disease and those having renal replacement therapy
* High use of inotropic and/or vasoactive agents at screening
* Electrocardiographic abnormalities
* Solid organ transplant recipient within 1 year of transplantation or one who presents with severe organ rejection

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2014-09-05 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (5):
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, München
- Novartis Investigative Site, Geneva, Switzerland
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 18 patients were assigned to study treatment. 6 patients were identified with GCP violations; hence, only 12 patients were included in disposition.
Groups:
- Serelaxin: Cohort 1: Serelaxin was administered intravenously on top of standard therapy for acute heart failure, for a total of 48 hours. In Cohort 1, patients in age group of 6 to <18 years were enrolled either into a low-dose or a high-dose group. During this 48-hour treatment period, the serelaxin dose rates to be administered were 3 μg/kg/day, 10 μg/kg/day and 30 μg/kg/day in the low -dose group; 10 μg/kg/day, 30 μg/kg/day and 100 μg/kg/day in the high-dose group. Both the low-dose and high- dose groups were planned to receive equal number of patients.
- Serelaxin: Cohort 2: Serelaxin was administered intravenously on top of standard therapy for acute heart failure, for a total of 48 hours. In Cohort 2, patients in age group of 1 to <6 years were enrolled either into a low-dose or a high-dose group. During this 48-hour treatment period, the serelaxin dose rates to be administered were 3 μg/kg/day, 10 μg/kg/day and 30 μg/kg/day in the low -dose group; 10 μg/kg/day, 30 μg/kg/day and 100 μg/kg/day in the high-dose group. Both the low-dose and high- dose groups were planned to receive equal number of patients.
- Serelaxin: Cohort 3: Serelaxin was administered intravenously on top of standard therapy for acute heart failure, for a total of 48 hours. In Cohort 3, patients in age group of 1 month to <1 year were enrolled either into a low-dose or a high-dose group. During this 48-hour treatment period, the serelaxin dose rates to be administered were 3 μg/kg/day, 10 μg/kg/day and 30 μg/kg/day in the low -dose group; 10 μg/kg/day, 30 μg/kg/day and 100 μg/kg/day in the high-dose group. In this cohort, high- dose group was planned to receive twice the number of patients in low-dose group.
Period: Overall Study
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Started | 8 | 3 | 1
Low-dose | 2 | 3 | 1
High-dose | 6 | 0 | 0
Completed | 8 | 3 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3 | Total
Number analyzed (Participants) | 8 | 3 | 1 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.1 (3.23) | 2.7 (1.53) | 0.7 (NA) — Standard Deviation cannot be calculated when there is one patient. | 8.1 (5.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 7 | 3 | 1 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 2 | 0 | 7
  Unknown or Not Reported | 3 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment Emergent Adverse Events, Serious Adverse Events and Death
Description: Number of patients with treatment emergent adverse events (including confirmed systolic blood pressure decreases and worsening heart failure), serious adverse events and death were reported.
Time Frame: through 28 days + 30 days SAE follow up after completion or discontinuation from the study
Population: All appropriately consented enrolled subjects who were exposed to study drug regardless of the exposure and have at least one post-baseline safety assessment.
Measure: Number; unit: Patients
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 8 | 3 | 1
Patients
  at least one Adverse Event | 6 | 3 | 0
  Serious Adverse Event | 3 | 1 | 0
  Death | 0 | 0 | 0

2. Primary Outcome: Pharmacokinetic Concentration for Low Dose 3-10-30 ug/kg/Day
Description: Pharmacokinetic (PK) concentration was presented as the surrogate for PK parameters, the original primary endpoint, due to the unavailability of the PK parameters Css and CL. Serelaxin concentration was determined in serum by a validated Enzyme Linked ImmunoSorbent Assay (ELISA) based upon the commercially available kit from R&D Systems (Catalogue No. DRL200). The ELISA method used a monoclonal antibody specific for human H2 relaxin as the capture reagent and an enzyme-linked polyclonal antibody specific for human.
Time Frame: at 0, 2, 16, 22, 32, 40, 48 hr. during the infusion, at 0.5, 4, 8 hours post infusion or study drug discontinuation, and on day 28
Population: participants with available data differed across time points
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 2 | 2 | 1
ng/mL
  Day 1 hour 0 during infusion | 0.083 (NA) — CV% geo-mean is derived as a function of log-transformed data. At least one patient had an outcome value = 0, causing the logarithm of the outcome value and thus CV% geo-mean undefined (note: logarithm of data can only be defined for a value > 0) | NA (NA) — All outcome value(s) = 0. Therefore, Geometric mean and CV% geo-mean are not populated. | NA (NA) — All outcome value(s) = 0. Therefore, Geometric mean and CV% geo-mean are not populated.
  Day 1 hour 2 during infusion | 0.514 (23.600) | 0.375 (176.043) | 1.250
  Day 1 hour 16 during infusion | 0.795 (66.578) | 0.772 (41.016) | 0.571
  Day 1 hour 22 during infusion | 2.868 (23.134) | 2.183 (11.690) | 3.810
  Day 2 hour 32 during infusion | 3.208 (32.740) | 2.155 (13.492) | NA (NA) — All outcome value(s) = 0. Therefore, Geometric mean and CV% geo-mean are not populated
  Day 2 hour 40 during infusion | 7.891 (49.702) | 5.513 (17.664) | 0.236
  Day 2 hour 48 during infusion | 6.315 (60.265) | 5.365 (16.148) | 9.010
  Day 3 hour 48.5 post infusion | 5.107 (39.153) | 3.999 (22.826) | 66.600
  Day 3 hour 52 post infusion | 1.751 (26.134) | 0.956 (12.016) | 2.440
  Day 3 hour 56 post infusion | 0.420 (42.285) | 0.416 (59.458) | 0.470
  Day28 hour 648 n=2,1,0 post infusion: number analyzed (Participants) | 2 | 1 | 0
  Day28 hour 648 n=2,1,0 post infusion | NA (NA) — All outcome value(s) = 0. Therefore, Geometric mean and CV% geo-mean are not populated | NA — All outcome value(s) = 0. Therefore, Geometric mean and CV% geo-mean are not populated |

3. Primary Outcome: Pharmacokinetic Concentration for High Dose (10-30-100 ug/kg/Day)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: No data available for Cohort 2 and 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 6 | 0 | 0
ng/mL
  Day 1 hour 0 during infusion | NA (NA) — At least one outcome value = 0. Geometric mean is calculated based on the logarithm of the outcome values, and is not populated if any outcome value = 0. CV is not available due to insufficient number of patients with measurement |  |
  Day 1 hour 2 during infusion: number analyzed (Participants) | 5 | 0 | 0
  Day 1 hour 2 during infusion | 2.388 (47.476) |  |
  Day 1 hour 16 during infusion | 4.004 (29.713) |  |
  Day 1 hour 22 during infusion: number analyzed (Participants) | 4 | 0 | 0
  Day 1 hour 22 during infusion | 9.774 (44.219) |  |
  Day 2 hour 32 during infusion: number analyzed (Participants) | 4 | 0 | 0
  Day 2 hour 32 during infusion | 10.472 (45.060) |  |
  Day 2 hour 40 during infusion: number analyzed (Participants) | 4 | 0 | 0
  Day 2 hour 40 during infusion | 35.515 (36.868) |  |
  Day 2 hour 48 during infusion: number analyzed (Participants) | 4 | 0 | 0
  Day 2 hour 48 during infusion | 39.777 (39.452) |  |
  Day 3 hour 48.5 post infusion: number analyzed (Participants) | 4 | 0 | 0
  Day 3 hour 48.5 post infusion | 27.818 (25.738) |  |
  Day 3 hour 52 post infusion: number analyzed (Participants) | 4 | 0 | 0
  Day 3 hour 52 post infusion | 7.014 (64.862) |  |
  Day 3 hour 56 post infusion: number analyzed (Participants) | 4 | 0 | 0
  Day 3 hour 56 post infusion | 2.576 (78.318) |  |
  Day 14 hour 312 post infusion: number analyzed (Participants) | 1 | 0 | 0
  Day 14 hour 312 post infusion | NA (NA) — At least one outcome value = 0. Geometric mean is calculated based on the logarithm of the outcome values, and is not populated if any outcome value=0.Geometric CV cannot be calculated due to insufficient number of participants with events |  |
  Day 28 hour 648 post infusion: number analyzed (Participants) | 3 | 0 | 0
  Day 28 hour 648 post infusion | NA (NA) — At least one outcome value = 0. Geometric mean is calculated based on the logarithm of the outcome values, and is not populated if any outcome value = 0. Geometric CV cannot be calculated due to insufficient number of participants with events |  |

4. Secondary Outcome: Change From Baseline in Mean Left Arterial Pressure for Low Dose (3-10-30 ug/kg/Day)
Description: The evaluations, as available, were done at baseline, prior to each dose escalation and at approximately 24 hours after the end of the infusion. Hemodynamic effects were also assessed for safety at additional time points during the study.
Time Frame: baseline, prior to each dose escalation, and at 24 hr. post end of infusion
Population: No data available
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in Mean Left Arterial Pressure for High Dose (10 -30-100 ug/kg/Day)
Description: as for outcome 4
Time Frame: baseline, prior to each dose escalation, and at 24 hr. post end of infusion
Population: No data available
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in Mean Pulmonary Artery Pressure (PAP- Systolic and Diastolic) for Low Dose (3-10-30 ug/kg/Day)
Description: The evaluations, as available, were done at baseline, prior to each dose escalation and at approximately 24 hours after the end of the infusion. Hemodynamic effects were also assessed for safety at additional time points during the study. Absolute values are presented at baseline; change from baseline values are presented at post-baseline time points
Time Frame: Day 1: hour 0 (Baseline) and 16, Day 2: hour 32 and 48, Day3: 24 hours post infusion
Population: participants with available data differed across time points
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 0 | 1 | 0
mmHg
  Baseline diastolic |  | 14.0 |
  Baseline systolic |  | 20.0 |
  Day 1 hour 16 diastolic |  | -2.0 |
  Day 1 hour 16 systolic |  | 3.0 |
  Day 2 hour 32 diastolic |  | 0.0 |
  Day 2 hour 32 systolic |  | -2.0 |
  Day 2 hour 48 diastolic |  | 11.0 |
  Day 2 hour 48 systolic |  | 6.0 |
  Day 3 24 hours post infusiondiastolic: number analyzed (Participants) | 0 | 0 | 0
  Day 3 24 hours post infusionsystolic: number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in Mean Pulmonary Artery Pressure (PAP- Systolic and Diastolic) for High Dose (10-30-100 ug/kg/Day)
Description: as for outcome 6
Time Frame: Day 1: hour 0 and 16, Day 2: hour 32 and 48, Day 3: 24 hours post infusion
Population: no data available for any time points
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Mean Central Venous Pressure for Low Dose (3-10-30 ug/kg/Day)
Description: as for outcome 6
Time Frame: Day 1: hour 0 (Baseline) and 16, Day 2: hour 32 and 48, Day 3: 24 hours post infusion
Population: participants with available data differed across time points
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 1 | 1 | 0
mmHg
  Baseline | 9.0 | 14.0 |
  Day 1 hour 16 | -1.0 | 2.0 |
  Day 2 hour 32: number analyzed (Participants) | 1 | 0 | 0
  Day 2 hour 32 | 2.0 |  |
  Day 2 hour 48: number analyzed (Participants) | 1 | 0 | 0
  Day 2 hour 48 | 2.0 |  |
  Day 3 24 hours post infusion: number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in Mean Central Venous Pressure for High Dose (10-30-100 ug/kg/Day)
Description: as for outcome 6
Time Frame: Day 1: hour 0 (Baseline) and 16, Day 2: hour 32 and 48, Day 3: 24 hours post infusion
Population: participants with available data differed across time points
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 1 | 0 | 0
mmHg
  Baseline | 4.0 |  |
  Day 1 hour 16 | 2.0 |  |
  Day 2 hour 32 | 3.0 |  |
  Day 2 hour 48 | 1.0 |  |
  Day 3 24 hours post infusion: number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Baseline and Change From Baseline in Mean Central Venous Pressure and Arterial Oxygen Saturation for Low Dose (3-10-30 ug/kg/Day)
Description: This analysis includes central venous and arterial oxygen saturation measurement, yielding a calculation of the arterio-venous oxygen extraction, where available at each time point. If no arterial access was available, then arterial oxygen saturation measurement data were obtained using a pulse oximeter. The evaluations, as available, were done at baseline, prior to each dose escalation and at approximately 24 hours after the end of the infusion. Hemodynamic effects were also assessed for safety at additional time points during the study. Absolute values are presented at baseline; change from baseline values are presented at post-baseline time points
Time Frame: Day 1: hour 0 (Baseline) and 16, Day 2: hour 32 and 48, Day 3: 24 hours post infusion
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 2 | 3 | 1
percentage of oxygen saturation
  Baseline | 99.5 (0.71) | 94.0 (6.56) | 100.0
  Day 1 our 16 | -4.5 (0.71) | -2.0 (3.00) | 0.0
  Day 2 hour 32 | -4.5 (2.12) | 1.3 (1.53) | -3.0
  Day 2 hour 48 | -3.0 (1.41) | -0.3 (1.53) | -2.0
  Day 3 - 24 hours post infusion | -5.0 (4.24) | 1.7 (1.53) | -3.0

11. Secondary Outcome: Baseline and Change From Baseline in Mean Central Venous Pressure and Arterial Oxygen Saturation for High Dose (10-30-100 ug/kg/Day)
Description: as for outcome 10
Time Frame: Day 1: hour 0 (Baseline) and 16, Day 2: hour 32 and 48, Day 3: 24 hours post infusion
Population: participants with available data differed across time points
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 6 | 0 | 0
percentage of oxygen saturation
  Baseline | 97.2 (2.56) |  |
  Day 1 our 16 | -0.2 (3.87) |  |
  Day 2 hour 32 | -0.2 (2.32) |  |
  Day 2 hour 48 | -0.2 (2.14) |  |
  Day 3 24 hours post infusion: number analyzed (Participants) | 5 | 0 | 0
  Day 3 24 hours post infusion | -0.2 (1.92) |  |

12. Secondary Outcome: Baseline and Change From Baseline in Mean Urine Output for Low Dose (3-10-30 ug/kg/Day)
Description: as for outcome 6
Time Frame: Day 1: hour 0 (Baseline) and 16, Day 2: hour 32 and 48, Day 3: 24 hours post infusion
Population: participants with available data differed across time points
Measure: Mean (Standard Deviation); unit: mL/kg/hour
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 2 | 3 | 1
mL/kg/hour
  Baseline: number analyzed (Participants) | 1 | 3 | 1
  Baseline | 2.0 | 1.3 (1.53) | 1.0
  Day 1 our 16: number analyzed (Participants) | 1 | 3 | 1
  Day 1 our 16 | -1.0 | 0.7 (1.15) | 0.0
  Day 2 hour 32: number analyzed (Participants) | 0 | 3 | 1
  Day 2 hour 32 |  | 3.7 (4.73) | -1.0
  Day 2 hour 48: number analyzed (Participants) | 0 | 3 | 1
  Day 2 hour 48 |  | 0.0 (2.00) | 0.0
  Day 3 24 hours post infusion: number analyzed (Participants) | 0 | 2 | 1
  Day 3 24 hours post infusion |  | 1.5 (2.12) | 0.0

13. Secondary Outcome: Baseline and Change From Baseline in Mean Urine Output for High Dose (10-30-100 ug/kg/Day)
Description: as for outcome 6
Time Frame: Day 1: hour 0 (Baseline) and 16, Day 2: hour 32 and 48, Day 3: 24 hours post infusion
Population: participants with available data differed across time points
Measure: Mean (Standard Deviation); unit: mL/kg/hour
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 6 | 0 | 0
mL/kg/hour
  Baseline | 2.2 (2.48) |  |
  Day 1 our 16: number analyzed (Participants) | 5 | 0 | 0
  Day 1 our 16 | -0.8 (2.59) |  |
  Day 2 hour 32: number analyzed (Participants) | 5 | 0 | 0
  Day 2 hour 32 | 0.0 (5.10) |  |
  Day 2 hour 48: number analyzed (Participants) | 5 | 0 | 0
  Day 2 hour 48 | -0.4 (2.70) |  |
  Day 3 24 hours post infusion: number analyzed (Participants) | 4 | 0 | 0
  Day 3 24 hours post infusion | -2.0 (2.71) |  |

14. Secondary Outcome: Baseline and Change From Baseline in Mean Blood Lactate Levels (Arterial Blood) for Low Dose (3-10-30 ug/kg/Day)
Description: as for outcome 6
Time Frame: Day 1: hour 0 (Baseline) and 16, Day 2: hour 32 and 48, Day 3: 24 hours post infusion
Population: participants with available data differed across time points
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 2 | 3 | 1
mmol/L
  Baseline: number analyzed (Participants) | 1 | 2 | 0
  Baseline | 3.900 | 2.560 (1.0748) |
  Day 1 our 16: number analyzed (Participants) | 1 | 1 | 0
  Day 1 our 16 | -3.100 | -0.500 |
  Day 2 hour 32: number analyzed (Participants) | 1 | 1 | 0
  Day 2 hour 32 | -3.100 | -1.100 |
  Day 2 hour 48: number analyzed (Participants) | 1 | 1 | 0
  Day 2 hour 48 | -3.200 | -0.900 |
  Day 3 24 hours post infusion: number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Baseline and Change From Baseline in Mean Blood Lactate Levels (Central Venous Blood) for Low Dose (3-10-30 ug/kg/Day)
Description: as for outcome 6
Time Frame: Day 1: hour 0 (Baseline) and 16, Day 2: hour 32 and 48, Day 3: 24 hours post infusion
Population: participants with available data differed across time points
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 2 | 3 | 1
mmol/L
  Baseline: number analyzed (Participants) | 1 | 1 | 0
  Baseline | 1.110 | 2.000 |
  Day 1 our 16: number analyzed (Participants) | 1 | 1 | 0
  Day 1 our 16 | 0.333 | 0 |
  Day 2 hour 32: number analyzed (Participants) | 1 | 0 | 0
  Day 2 hour 32 | -0.222 |  |
  Day 2 hour 48: number analyzed (Participants) | 1 | 1 | 0
  Day 2 hour 48 | 0.111 | 0 |
  Day 3 24 hours post infusion: number analyzed (Participants) | 1 | 0 | 0
  Day 3 24 hours post infusion | -0.222 (NA) — Standard deviation cannot be calculated due to insufficient number of patients with measurement |  |

16. Secondary Outcome: Baseline and Change From Baseline in Mean Blood Lactate Levels (Arterial Blood) for High Dose (10-30-100 ug/kg/Day)
Description: as for outcome 6
Time Frame: Day 1: hour 0 (Baseline) and 16, Day 2: hour 32 and 48, Day 3: 24 hours post infusion
Population: participants with available data differed across time points
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 1 | 0 | 0
mmol/L
  Baseline | 1.300 |  |
  Day 1 our 16 | -0.100 |  |
  Day 2 hour 32 | 0.200 |  |
  Day 2 hour 48 | -0.300 |  |
  Day 3 24 hours post infusion: number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Baseline and Change From Baseline in Mean Blood Lactate Levels (Central Venous Blood) for High Dose (10-30-100 ug/kg/Day)
Description: as for outcome 6
Time Frame: Day 1: hour 0 (Baseline) and 16, Day 2: hour 32 and 48, Day 3: 24 hours post infusion
Population: participants with available data differed across time points
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
Number analyzed (Participants) | 2 | 0 | 0
mmol/L
  Baseline: number analyzed (Participants) | 1 | 0 | 0
  Baseline | 1.200 |  |
  Day 1 our 16: number analyzed (Participants) | 1 | 0 | 0
  Day 1 our 16 | -0.600 (NA) — Standard deviation cannot be calculated due to insufficient number of patients with measurement |  |
  Day 2 hour 32: number analyzed (Participants) | 0 | 0 | 0
  Day 2 hour 48: number analyzed (Participants) | 1 | 0 | 0
  Day 2 hour 48 | -0.200 (NA) — Not available due to insufficient number of patients with measurement |  |
  Day 3 24 hours post infusion: number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected for the maximum actual duration of treatment exposure and follow-up (i.e. approximately 28 days) for the participants per protocol
Arm/Group | Serelaxin: Cohort 1 | Serelaxin: Cohort 2 | Serelaxin: Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 3/8 | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 6/8 | 3/3 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Serelaxin: Cohort 1 (N=8) | Serelaxin: Cohort 2 (N=3) | Serelaxin: Cohort 3 (N=1)
Atrial thrombosis (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Serelaxin: Cohort 1 (N=8) | Serelaxin: Cohort 2 (N=3) | Serelaxin: Cohort 3 (N=1)
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood pressure systolic decreased (Investigations) | 1 | 0 | 0
Cardioactive drug level increased (Investigations) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin oedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, the planned analyses were not performed as the limited set of data would preclude meaningful interpretation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT02151383/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT02151383/SAP_001.pdf